CLINICAL TRIAL: NCT05273437
Title: Control Systems Engineering for Counteracting Notification Fatigue: An Examination of Health Behavior Change.
Brief Title: The JustWalk JITAI Study: A System Identification Experiment to Understand Just-in-Time States of Physical Activity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: National Library of Medicine (NLM) (NIH)
Responsible Party: Principal Investigator, Eric Hekler, Professor, University of California, San Diego
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 800132; 5R01LM013107 (NIH)
Record Dates: First submitted 2022-02-22; First posted 2022-03-10 (Actual); Results first posted 2024-11-19 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-10

CONDITIONS: Physical Inactivity; Health Behavior; Healthy Lifestyle
MeSH Terms: conditions — Sedentary Behavior; Health Behavior | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: See study description for details. All participants will receive all intervention elements, with provision varying across time experimentally using procedures appropriate for system identification.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- System Identification (Experimental): All participants in the study will go through a system identification experiment everyday for 270 days.
  Interventions: Behavioral: System identification experiment for physical activity

INTERVENTIONS:
Behavioral: System identification experiment for physical activity — The system identification experiment in Just Walk JITAI study has two key components that are the focus of the system identification experiment: daily adaptive step goal recommendations and within-day suggestions to either plan a bout of walking or to inspire reflection and, by extension, an increased urge to go for a walk.

SUMMARY:
The goal of this system identification experiment is to estimate and validate dynamical computational models that can be used in a future a multi-timescale model-predictive controller. System identification is an experimental approach used in control systems engineering, which uses random and pseudo-random signal designs to experimentally manipulate independent variables, with the goal of producing dynamical models that can meaningfully predict individual responses to varying provision of support. A system identification is single subject/N-of-1 experimental design, whereby each person is their own control. This 9-month system identification experiment will experimentally vary daily suggested step goals and provision of notifications meant to inspire bouts of walking during different plausible just-in-time states. Results of this system identification experiment will then enable the development a future multi-timescale model-predictive controller-driven just-in-time adaptive intervention (JITAI) intended to increase steps/day. The system identification experiment will be conducted among N=50 inactive, adults aged 21 or over who have no preexisting conditions that preclude them from engaging in an exercise program, as determined using the physical activity readiness questionnaire.

DETAILED DESCRIPTION:
N=50 English-speaking adults aged 21+ who are physically inactive (self-reported engagement in less than 60 minutes/week of moderate-intensity activity) and own a smartphone (iPhone or Android) will be recruited. Participants will be provided with and asked to wear a Fitbit Versa 3 and use the study app, JustWalk, for 270 days.

A system identification experiment, which is a single subject/N-of-1 experimental protocol used in control systems engineering, will be conducted. This study is designed to empirically optimize dynamical models that can be used within a future model-predictive controller-driven just-in-time adaptive intervention (JITAI). This system identification experiment will include two experimentally manipulated components: 1) notifications delivered up to 4 time per day designed to increase a person's steps within the next 3 hours via either increased awareness of the urge to walk or via bout planning; and 2) adaptive daily step goal suggestions. Both components will be experimentally manipulated using procedures appropriate for system identification. Specifically, notifications prompting planning of short walks within the next 3 hours will be experimentally provided or not across variations of need (i.e., whether daily step goals were previously met), opportunity (i.e., the next three hours is a time window when a person previously walked), and receptivity (i.e., person received fewer than 6 messages in the last 72 hours and walked after notifications were sent). This enables experimental manipulation of varying "just-in-time" states, thus providing valuable data for guiding future predictions about when, where, and for whom a bout notification would produce the desired effects compared to not. Thus, this is a hypothesis-driven approach to better understanding issues of notification fatigue by seeking to provide notifications only when said notifications are needed, when a person has the opportunity to act on them, and is receptive to receiving support. In addition, suggested daily step goals will also be varied systematically across time. A suggested step goal will vary between a person's median steps/day, calculated from the person's previous activity measured via Fitbit, up to 3,000 steps above their median reference. The goals will continue to get progressively more difficult if a person meets their suggested step goals. The system will stop increasing suggested step goals if a person achieves a median of 12,000 steps/day as their reference. During the study, participants will wear a Fitbit for the duration to measure PA and also fill out ecological momentary assessment surveys of psychological constructs hypothesized to be key variables for the targeted dynamical computational models.

After study completion, dynamical modeling analyses appropriate for system identification will be conducted for each participant (see references for more details on the types of analyses that will be conducted). The goal is to estimate and validate the dynamical computational models, with a particular benchmark used on the degree to which a dynamical model can predict, prospectively, each person's future steps/day and response to a particular bout notification. Results from this dynamical systems modeling will then enable the development of a multi-timescale model-predictive controller driven JITAI designed to provide support for increasing walking among healthy adults, which can then be tested in a future clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* inactive: engaging in less than 60 min/week of self-reported moderate intensity physical activity
* adults: aged 21 or older
* own a smartphone that can run HeartSteps (iOS or Android)

Exclusion Criteria:

* not proficient in English, or
* indicate medical problems that preclude physical activity as defined using physical activity readiness questionnaire (PAR-Q)

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-04-11 (Actual); Primary Completion 2023-05-15 (Actual); Study Completion 2023-05-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Hekler, PhD, Principal Investigator — University of California, San Diego
Locations (1):
- University of California San Diego, San Diego, California, United States

REFERENCES:
- [Background] Hekler EB, Rivera DE, Martin CA, Phatak SS, Freigoun MT, Korinek E, Klasnja P, Adams MA, Buman MP. Tutorial for Using Control Systems Engineering to Optimize Adaptive Mobile Health Interventions. J Med Internet Res. 2018 Jun 28;20(6):e214. doi: 10.2196/jmir.8622. PMID 29954725
- [Background] Phatak SS, Freigoun MT, Martin CA, Rivera DE, Korinek EV, Adams MA, Buman MP, Klasnja P, Hekler EB. Modeling individual differences: A case study of the application of system identification for personalizing a physical activity intervention. J Biomed Inform. 2018 Mar;79:82-97. doi: 10.1016/j.jbi.2018.01.010. Epub 2018 Feb 1. PMID 29409750
- [Background] Korinek EV, Phatak SS, Martin CA, Freigoun MT, Rivera DE, Adams MA, Klasnja P, Buman MP, Hekler EB. Adaptive step goals and rewards: a longitudinal growth model of daily steps for a smartphone-based walking intervention. J Behav Med. 2018 Feb;41(1):74-86. doi: 10.1007/s10865-017-9878-3. Epub 2017 Sep 16. PMID 28918547
- [Derived] Park J, Kim M, El Mistiri M, Kha R, Banerjee S, Gotzian L, Chevance G, Rivera DE, Klasnja P, Hekler E. Advancing Understanding of Just-in-Time States for Supporting Physical Activity (Project JustWalk JITAI): Protocol for a System ID Study of Just-in-Time Adaptive Interventions. JMIR Res Protoc. 2023 Sep 26;12:e52161. doi: 10.2196/52161. PMID 37751237

RESULTS

PARTICIPANT FLOW:
Groups:
- System Identification: All participants in the study will go through a system identification experiment everyday for 270 days. System identification experiment for physical activity: The system identification experiment in Just Walk JITAI study has two key components that are the focus of the system identification experiment: walking suggestions and daily step goals. To achieve the desired dynamics on the timescale of interest, we used 2 input signals, one for each of the 2 components. Although our study design enables traditional statistical analyses to examine the impact of intervention components on behavioral outcomes, that is not the primary focus of a system ID experiment. The primary goal of a system ID experiment is to estimate and validate dynamical computational models that are validated based on their ability to predict the future responses of each individual's behavior across time. These aims are achieved by having different intervention components-suggestions to walk in the next 3 hours and adaptive goal setting-delivered at different timescales and orthogonally, that is, statistically independent of each other.
Period: Overall Study
Arm/Group | System Identification
Started | 50
Completed | 48
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | System Identification
Number analyzed (Participants) | 48
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 48
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.4 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: There were 3 missing data for this measure.
  Participants
    number analyzed (Participants) | 45
    Female | 29
    Male | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: There were 3 missing data for this measure.
  Participants
    number analyzed (Participants) | 45
    Hispanic or Latino | 8
    Not Hispanic or Latino | 37
    Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: There were 4 missing data for this measure.
  Participants
    number analyzed (Participants) | 44
    American Indian or Alaska Native | 1
    Asian | 14
    Native Hawaiian or Other Pacific Islander | 3
    Black or African American | 2
    White | 17
    More than one race | 2
    Unknown or Not Reported | 5
Region of Enrollment [Number; unit: participants]
  United States | 48

OUTCOME MEASURES:

1. Primary Outcome: Steps/Day
Description: This will be measured continuously for the duration of the study via a Fitbit Versa, a wrist-worn, consumer-level activity tracker.
Time Frame: Everyday from baseline to the end of study (for 270 days)
Measure: Number; unit: Steps/day
Arm/Group | System Identification
Number analyzed (Participants) | 44
Steps/day
  Participant 1 | 4048.4
  Participant 2 | 1074.4
  Participant 3 | 1645.8
  Participant 4 | 1749.1
  Participant 5 | 2991.3
  Participant 6 | NA — Daily intervention effect on Weekend is not available.
  Participant 7 | 1254.6
  Participant 8 | 2168.3
  Participant 9 | 1471.5
  Participant 10 | 2003.8
  Participant 11 | NA — Daily intervention effect on both Weekday and Weekend are not available.
  Participant 12 | 1333.0
  Participant 13 | 1168.5
  Participant 14 | 2577.2
  Participant 15 | 2703.3
  Participant 16 | 1819.4
  Participant 17 | 1930.3
  Participant 18 | 2229.0
  Participant 19 | 295.0
  Participant 20 | 1887.8
  Participant 21 | 1563.3
  Participant 22 | 704.9
  Participant 23 | 1703.3
  Participant 24 | 156.4
  Participant 25 | 1187.5
  Participant 26 | 3697.9
  Participant 27 | 1138.1
  Participant 28 | 1470.2
  Participant 29 | 919.0
  Participant 30 | NA — Daily intervention effect on both Weekday and Weekend are not available.
  Participant 31 | 1015.9
  Participant 32 | NA — Daily intervention effect on both Weekday and Weekend are not available.
  Participant 33 | 449.8
  Participant 34 | 1228.2
  Participant 35 | 1074.1
  Participant 36 | 967.1
  Participant 37 | 2928.6
  Participant 38 | 2608.3
  Participant 39 | 738.2
  Participant 40 | 2677.5
  Participant 41 | 783.5
  Participant 42 | 1631.8
  Participant 43 | 1387.4
  Participant 44 | 1008.3
Statistical Analysis 1: Comparison: System Identification; We hypothesized that some individuals have their own time and decision-policy-specific response pattern regardless of day elapsed since the beginning of the intervention. We did not hypothesize the direction of the effect variation; Test type: Other — We conducted a Bayesian Regression for all available participants, then visualized the results. (N x 16 table, N: number of participants); Bayesian Regression; We explicitly sought 80% credibility of at least 100 steps more within the 3-hour increment in comparison to the intervention; Credibility interval = 80 — We decided that 100 steps/3 hours is the minimum value of the MAP intervention effect estimate and that an INUS condition is valid only if there is at least an 80% chance of achieving an effect beyond 100 steps/3 hours; The decision point was the unit of analysis. For the Bayesian Regression, we used Markov Chain Monte Carlo (MCMC). Four sampling chains were used when performing Bayesian modeling. The number of estimation samples and target acceptance rate were gradually increased until numerical stability was achieved. The number of estimation samples was increased by multiplied by 2, as advised by previous literature, depending on the ratio of convergence diagnostics R̂ > 1.1. We used 100 steps increase during 3 hours as the effect threshold value. We assumed that there is an effect only if the estimated effect is more than 80% probable (i.e., the credibility interval is over 100 steps/3 hours) and the Maximum A Posteriori Point (MAP) of the effect is more than 100 steps/3 hours. Otherwise, there is no effect. Among the models with effects, we clipped to 1000 steps/3hours as a maximum if the MAP was greater than 1000 steps/3 hours

ADVERSE EVENTS:
Time Frame: The adverse event data were collected from the enrollment period to the end of intervention period which was about 10 months.
Description: Walking, even if it is a voluntary activity, may produce light-headedness, fatigue, or chest discomfort, especially under severe weather. There is also a risk of a cardiac event, such as a heart attack. This risk is less than 1 occurrence in 12,000 maximal exercise tests on healthy participants, and approximately 1-2 occurrences in 10,000 maximal tests on higher risk participants. The risks involved in this study are no more than minimal.
Groups:
- System Identification: In the intervention phase, all app features were delivered, including the 2 push intervention components (ie, walking prompts and adaptive suggested step goals) and the daily EMA questions. The participants also gained access to other parts of the JustWalk JITAI app such as activity logs and planning support. Participants were asked to interact with the app whenever it sent them notifications and were told that they could open the app at any time if they wanted to access pull components and found them useful. Total interaction time with the app from push interventions and EMA notifications does not exceed 10 minutes each day, but participants may choose to spend more time on the app accessing other features.
Arm/Group | System Identification
All-Cause Mortality (participants affected / at risk) | 0/50
Serious Adverse Events (participants affected / at risk) | 0/50
Other Adverse Events (participants affected / at risk) | 0/50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-01-12): https://cdn.clinicaltrials.gov/large-docs/37/NCT05273437/Prot_SAP_002.pdf
  • Informed Consent Form (2022-01-12): https://cdn.clinicaltrials.gov/large-docs/37/NCT05273437/ICF_001.pdf